CLINICAL TRIAL: NCT01877577
Title: Supplementation of Vitamin D3 (Cholecalciferol) in Patients With Inflammatory Bowel Diseases (IBD) and Hypovitaminosis D: A Prospective Randomized Controlled Trial.
Brief Title: Supplementation of Vitamin D3 in Patients With Inflammatory Bowel Diseases and Hypovitaminosis D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IBDVitD-42012
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Crohn's Disease (CD); Ulcerative Colitis (UC)
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2000 I/U Vitamin D3 (Active Comparator): 2000 I/U Vitamin D3 Daily
  Interventions: Dietary Supplement: Vitamin D3
- 4000 I/U Vitamin D3 (Active Comparator): 4000 I/U Vitamin D3 Daily
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Study patients who took 2,000 IU daily of vitamin D3 will be compared to those who took 4,000 IU daily to determine the different effects of vitamin D3 dose on quality of life, disease activity, and the laboratory tests in this study.
  Other Names: vitamin D3 cholecalciferol

SUMMARY:
This study aims to evaluate the effect of vitamin D3 supplementation on disease activity and quality of life in IBD patients deficient in vitamin D, and also help determine the optimal dose of vitamin D3 for them.

Hypothesis: Supplementation of vitamin D3 in IBD patients with hypovitaminosis D can improve their quality of life and decrease IBD activity.

DETAILED DESCRIPTION:
The incidence of hypovitaminosis D has been reported to be as high as 75% in patients with IBD. However, it is unclear whether low vitamin D levels contribute to the pathogenesis of IBD or are a consequence of IBD. Recent animal data studies suggest that maintenance of the epithelial barrier integrity in the large intestine by vitamin D is important in preventing IBD.

However, more evidence is required to determine the effect of vitamin D3 supplementation in patients with IBD. Furthermore, there is no clear consensus regarding the appropriate dose of vitamin D supplementation in IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease (Crohn's disease, ulcerative colitis)
* 18 years of age or older
* 25(OH)D levels <30ng/ml
* willing to give informed written consent

Exclusion Criteria:

* Age < 18 years
* Women who are pregnant or planning to become pregnant
* Patients already taking vitamin D3 ≥2,000 IU/daily prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
vitamin D3 supplementation in IBD patients with hypovitaminosis D. | 90 days after patient taking the Vitamin D3 supplement daily
  To determine the appropriate dose of vitamin D3 supplementation in IBD patients with hypovitaminosis D.

SECONDARY OUTCOMES:
vitamin D3 supplementation on disease activity and quality of life | 90 days after patient taking the Vitamin D3 supplement daily
  To assess the effect of vitamin D3 supplementation on IBD disease activity and quality of life in patients with IBD and hypovitaminosis D.

CONTACTS AND LOCATIONS:
Overall Officials: David Limsui, MD, Principal Investigator — Assistant Clinical Professor, UCSF
Locations (1):
- Community Regional Medical Center, Ambulatory Care Center, Fresno, California, United States

REFERENCES:
- [Background] Khor B, Gardet A, Xavier RJ. Genetics and pathogenesis of inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):307-17. doi: 10.1038/nature10209. PMID 21677747
- [Background] Ulitsky A, Ananthakrishnan AN, Naik A, Skaros S, Zadvornova Y, Binion DG, Issa M. Vitamin D deficiency in patients with inflammatory bowel disease: association with disease activity and quality of life. JPEN J Parenter Enteral Nutr. 2011 May;35(3):308-16. doi: 10.1177/0148607110381267. PMID 21527593
- [Background] Kong J, Zhang Z, Musch MW, Ning G, Sun J, Hart J, Bissonnette M, Li YC. Novel role of the vitamin D receptor in maintaining the integrity of the intestinal mucosal barrier. Am J Physiol Gastrointest Liver Physiol. 2008 Jan;294(1):G208-16. doi: 10.1152/ajpgi.00398.2007. Epub 2007 Oct 25. PMID 17962355
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827